CLINICAL TRIAL: NCT00553761
Title: Pattern Electroretinogram and Multifocal Pattern Electroretinogram For the Detection of Neural Loss in Patients With Permanent Temporal Visual Field Defect From Chiasmal Compression
Brief Title: PERG and mfPERG in Band Atrophy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Mario Luiz Ribeiro Monteiro/University of Sao Paulo, University of Sao Paulo
Other Study IDs: 654/06; FAPESP 06/61549-6; 07/54142-0)
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2007-11

CONDITIONS: Band Atrophy
Keywords: Band atrophy; Pattern electroretinogram; Chiasmal compression; Neural loss; Electrophysiological tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pattern electroretinogram — Full field and hemifield (nasal and temporal) stimulation transient pattern electroretinogram (PERG) were recorded both in patients and controls.

SUMMARY:
The study is designed to evaluate the ability of pattern electroretinogram (PERG) and multifocal pattern electroretinogram (mfPERG) to measure and identify the pattern of band atrophy of the optic nerve in patients with long standing chiasmal lesions. The hypothesis is that these electrophysiological tests were able to identify this such pattern. The idea is to investigate the ability of the these electrophysiological technics in detecting the neural loss from chiasmal compression and to evaluate the ability of PERG and mfPERG parameters to differentiate between eyes with band atrophy of the optic nerve and healthy eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Visual acuity better than 20/30
2. Refractive error less 5 spherical diopter and 3 cylinder diopter
3. Temporal field defect

Exclusion Criteria:

1. Presence of glaucoma and optic nerve anomalies
2. Anormal nasal field

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with band atrophy from chismal compression and controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mário Luiz R Monteiro, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Monteiro ML, Hokazono K, Cunha LP, Oyamada MK. Correlation between multifocal pattern electroretinography and Fourier-domain OCT in eyes with temporal hemianopia from chiasmal compression. Graefes Arch Clin Exp Ophthalmol. 2013 Mar;251(3):903-15. doi: 10.1007/s00417-012-2156-8. Epub 2012 Sep 29. PMID 23052713
- [Derived] Monteiro ML, Hokazono K, Cunha LP, Oyamada MK. Multifocal pattern electroretinography for the detection of neural loss in eyes with permanent temporal hemianopia or quadrantanopia from chiasmal compression. Br J Ophthalmol. 2012 Jan;96(1):104-9. doi: 10.1136/bjo.2010.199661. Epub 2011 Mar 17. PMID 21415059
- [Derived] Monteiro ML, Cunha LP, Costa-Cunha LV, Maia OO Jr, Oyamada MK. Relationship between optical coherence tomography, pattern electroretinogram and automated perimetry in eyes with temporal hemianopia from chiasmal compression. Invest Ophthalmol Vis Sci. 2009 Aug;50(8):3535-41. doi: 10.1167/iovs.08-3093. Epub 2009 Mar 5. PMID 19264884
- [Derived] Cunha LP, Oyamada MK, Monteiro ML. Pattern electroretinograms for the detection of neural loss in patients with permanent temporal visual field defect from chiasmal compression. Doc Ophthalmol. 2008 Nov;117(3):223-32. doi: 10.1007/s10633-008-9126-9. Epub 2008 Apr 10. PMID 18401605
- See also: Pattern Electroretinograms For the Detection of Neural Loss in Patients with Permanent Temporal Visual Field Defect from Chiasmal Compression — http://www.ncbi.nlm.nih.gov/sites/entrez